CLINICAL TRIAL: NCT05067231
Title: UAB Cardiovascular Research Biobank
Brief Title: CARBON: UAB Cardiovascular Research Biobank
Acronym: CARBON
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pankaj Arora, MD, Assistant Professor, Division of Cardiovascular Disease, Department of Medicine, University of Alabama at Birmingham
Other Study IDs: IRB - 300007834
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Natriuretic Peptides; Cardiovascular Diseases; Hypertension; Diabetes; Obesity
Keywords: Natriuretic Peptides; Cardiovascular Diseases; Hypertension; Diabetes; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA, Plasma and Serum to be collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The UAB Cardiovascular Research Biobank (CARBON) will be a resource that contains biological materials, such as DNA samples, in addition to health and personal information on a large number of people over time. It will be set up so that it can be used in the future as a resource for researchers undertaking a wide range of medical research.

DETAILED DESCRIPTION:
The UAB Cardiovascular Research Biobank (CARBON) will be a resource that contains pertinent genetic, health, and biological samples such as blood derived from a large-scale population. Researchers may use disease correlates and predictors identified from the genetic, health, and personal information contained in the Biobank as a resource to investigate cardiovascular disease, hypertension, diabetes, and a myriad of other disorders. Through these studies, researchers may identify the progression of risk factors in certain diseases and help develop novel strategies to detect, treat, or prevent such diseases. In addition, the Biobank serves as a valuable tool to assess how certain treatments may respond differently to individuals as a result of genotypic differences.

The investigators have demonstrated that lower natriuretic peptide (NP) levels are associated with a decreased insulin sensitivity and have a causal role in the development of diabetes and have also shown that certain populations, such as African Americans, have relatively low NP levels, which may contribute to their underlying risk for insulin resistance. Since NPs play an important role in the regulation of insulin sensitivity, one can infer that relatively low NP levels are an important biological contributor to the high prevalence rates of cardiometabolic disease in African Americans. The Biobank will contain genetic information concerning the presence of gene variants that encode NPs.

ELIGIBILITY:
Inclusion Criteria:

* Age more than or equal to 18

Exclusion Criteria:

* Age <18, at screening
* Employees or students associated with the Division of Cardiovascular Disease at UAB will not be recruited due to their vulnerable status and susceptibility to coercion.
* Women who are pregnant or who can become pregnant and not practicing an acceptable method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals living in the Birmingham area will be enrolled through the University of Alabama at Birmingham campus. We will also enroll individuals who are associated with the University of Alabama at Birmingham.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Genetic Variants in the NPPA and NPPB gene of the Natriuretic Peptide family associated with the Cardiovascular and Metabolic Diseases | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Arora, MD, FAHA, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bajaj NS, Gutierrez OM, Arora G, Judd SE, Patel N, Bennett A, Prabhu SD, Howard G, Howard VJ, Cushman M, Arora P. Racial Differences in Plasma Levels of N-Terminal Pro-B-Type Natriuretic Peptide and Outcomes: The Reasons for Geographic and Racial Differences in Stroke (REGARDS) Study. JAMA Cardiol. 2018 Jan 1;3(1):11-17. doi: 10.1001/jamacardio.2017.4207. PMID 29167879